CLINICAL TRIAL: NCT07125846
Title: Clinical, Radiographic and Histologic Assessment of the Efficacy of Bioactive Glass as a Novel Grafting Material in Maxillary Sinus Floor Augmentation: A Randomized Controlled Study
Brief Title: Efficacy of Bioactive Glass vs. Xenograft in Maxillary Sinus Augmentation
Acronym: BIOXENO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MF-SINUS-2025
Record Dates: First submitted 2025-07-14; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Alveolar Bone Loss; Maxillary Sinus Disease; Tooth Loss
Keywords: Maxillary Sinus Augmentation; Bioactive Glass; Xenograft; Sinus Lift; Bone Grafting; Dental Implant
MeSH Terms: conditions — Alveolar Bone Loss; Tooth Loss

STUDY DESIGN:
Intervention Model Description: Two-arm parallel randomized controlled trial with 1:1 allocation ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioactive Glass Group (Experimental): Patients in this group will undergo maxillary sinus floor augmentation using bioactive glass bone graft material (UNIGRAFT, Biomed Inc., USA). The procedure will be performed via open sinus lift approach.
  Interventions: Device: Bioactive Glass Bone Graft (UNIGRAFT)
- Xenograft Group (Active Comparator): Patients in this group will undergo maxillary sinus floor augmentation using a conventional xenograft material via open sinus lift approach.
  Interventions: Device: Xenograft Bone Graft (Bio-Oss)

INTERVENTIONS:
Device: Bioactive Glass Bone Graft (UNIGRAFT) — A bioactive glass bone graft material (UNIGRAFT, Biomed Inc., USA) used for maxillary sinus floor augmentation via open sinus lift technique.
  Arms: Bioactive Glass Group
Device: Xenograft Bone Graft (Bio-Oss) — A commercially available bovine-derived xenograft material (Bio-Oss, Geistlich Pharma) used for maxillary sinus floor augmentation via open sinus lift technique.
  Arms: Xenograft Group

SUMMARY:
This randomized controlled study aims to evaluate the clinical, radiographic, and histologic efficacy of using bioactive glass bone graft (UNIGRAFT by Biomed Inc., USA) compared to a conventional xenograft in maxillary sinus augmentation procedures. A total of 20 patients classified as SA4 according to the Misch classification will be enrolled and randomly allocated into two groups. Outcomes will be assessed using Cone Beam Computed Tomography (CBCT) for vertical bone gain and, where applicable, histologic analysis. The study is conducted at the Faculty of Dentistry, Suez Canal University.

DETAILED DESCRIPTION:
The aim of this clinical study is to compare the performance of a novel bioactive glass bone graft (UNIGRAFT) with a standard xenograft material in open sinus lift procedures for patients with severely atrophic maxillary posterior ridges (Misch SA4 classification). The trial is designed as a parallel-arm, randomized controlled study involving 20 patients. Each participant will undergo maxillary sinus augmentation using either the bioactive glass or the xenograft, followed by a healing period prior to implant placement.

Radiographic evaluation using CBCT will be conducted to assess vertical bone height gain pre- and post-operatively. Additionally, histological samples may be obtained during implant placement in indicated cases to evaluate bone quality. The primary endpoint is vertical bone gain after 6 months, and secondary endpoints include bone density, complication rate, and histologic characteristics. The study will follow strict ethical guidelines and is approved by the institutional ethics committee of Suez Canal University.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring maxillary sinus floor augmentation for dental implant placement.
* Residual alveolar bone height ≤ 4 mm in posterior maxilla (SA4 classification).
* Age between 20 to 65 years.
* Good general health and able to attend scheduled follow-up visits.
* Signed written informed consent.

Exclusion Criteria:

* Presence of systemic conditions that could affect bone healing (e.g., uncontrolled diabetes, osteoporosis).

History of radiotherapy in the head and neck region.

* Heavy smoking (more than 10 cigarettes/day).
* Active sinus pathology or previous sinus surgery.
* Pregnant or breastfeeding women.
* Use of medications affecting bone metabolism (e.g., bisphosphonates or corticosteroids).
* Poor oral hygiene or untreated periodontal disease.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in vertical bone height measured by CBCT | 6 months after sinus augmentation
  Evaluation of the change in vertical bone height in the grafted sinus area using CBCT imaging. CBCT scans will be taken preoperatively and at 6 months postoperatively to assess bone formation

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Elsholkamy, Professor, Principal Investigator — Suez Canal University

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results of the study may be shared publicly or upon request after publication. Data sharing will be at the discretion of the principal investigator and will not require prior approval from external parties. The data will be used solely for academic and non-commercial purposes.
Supporting Information: SAP, ICF
Time Frame: Data will be available beginning 6 months after the primary completion date and will be accessible for up to 3 years.
Access Criteria: Qualified researchers may request access to the de-identified data by contacting the principal investigator. Access will be granted for academic purposes only. A data use agreement may be required.

REFERENCES:
- [Background] Cordioli G, Mazzocco C, Schepers E, Brugnolo E, Majzoub Z. Maxillary sinus floor augmentation using bioactive glass granules and autogenous bone with simultaneous implant placement. Clinical and histological findings. Clin Oral Implants Res. 2001 Jun;12(3):270-8. doi: 10.1034/j.1600-0501.2001.012003270.x. PMID 11359485
- [Background] Pereira RS, Menezes JD, Bonardi JP, Griza GL, Okamoto R, Hochuli-Vieira E. Comparative study of volumetric changes and trabecular microarchitecture in human maxillary sinus bone augmentation with bioactive glass and autogenous bone graft: a prospective and randomized assessment. Int J Oral Maxillofac Surg. 2018 May;47(5):665-671. doi: 10.1016/j.ijom.2017.11.016. Epub 2017 Dec 13. PMID 29246424
- See also: Official product page for Unigraft® bioactive glass synthetic bone graft used in maxillary sinus augmentation procedures. — https://www.unicarebiomedical.com/dental-supplies/unigraft.html

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-06-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT07125846/Prot_SAP_ICF_000.pdf